CLINICAL TRIAL: NCT04827680
Title: Clinical Evaluation of the Safety and Performance of Fractional Radiofrequency for the Treatment and Reduction of Acne Scarring
Brief Title: Clinical Evaluation of the Safety and Performance of FRF for the Treatment and Reduction of Acne Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VI0121
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
Keywords: acne scarring; acne scar; fractional radiofrequency; fractional RF; FRF
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Masking Description: Blinded evaluation of photographs taken at baseline and at 6, 12 weeks post final treatment by independent evaluators.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All subjects (Experimental): The Venus Viva™ fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids and scars. Beginning with the Baseline visit (Visit 1), subjects will receive a total of 3 treatments approximately 3-5 weeks apart.
  Interventions: Device: Venus Viva MD

INTERVENTIONS:
Device: Venus Viva MD — The Venus Viva™ MD fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids, and scars. Beginning with the Baseline visit (Visit 1), subjects will receive a total of 3 treatments approximately 3-5 weeks apart.

SUMMARY:
Prospective, single centre, evaluator-blind study of the safety and performance of fractional radiofrequency (RF) for the treatment and reduction of acne scarring. The study will evaluate the progress of 20 subjects requesting treatment of acne scarring. The study will involve three treatments on both sides of the face with 3-5 week intervals between each treatment. Subjects will be followed at 6 and 12 weeks after their last treatment. Analysis will be performed on all subjects who receive at least one treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subjects over 21 years of age who are seeking treatment and reduction of their acne scarring.
2. Able to read, understand and voluntarily provide written Informed Consent.
3. Able and willing to comply with the treatment/follow-up schedule and requirements.
4. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study and have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

1. Implantable defibrillators, cardiac pacemakers, and other metal implants
2. Subjects with any implantable metal device in the treatment area
3. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body (e.g. cochlear implant).
4. Permanent implant in the treated area, such as metal plates and screws, or an injected chemical substance.
5. Current or history of any kind of cancer, or pre-malignant moles.
6. Severe concurrent conditions, such as cardiac disorders.
7. Pregnancy or intending to become pregnant during the study and nursing.
8. Impaired immune system due to immunosuppressive diseases, such as AIDS and HIV, or use of immunosuppressive medications.
9. History of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area; may be enrolled only after a prophylactic regime has been followed for 2 weeks or longer prior to enrollment, or according to Investigator's discretion.
10. Poorly controlled endocrine disorders, such as diabetes.
11. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
12. History of skin disorders, such as keloids, abnormal wound healing, as well as very dry and fragile skin.
13. History of bleeding coagulopathies, or use of anticoagulants (excluding daily aspirin).
14. Facial dermabrasion, facial resurfacing, or deep chemical peeling within the last three months, if face is treated.
15. Use of isotretinoin (Accutane®) or other systemic retinoids within six months or topical retinoids within three months prior to treatment; or as per physician's discretion.
16. Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g. ibuprofen containing agents) one week before and after each treatment session.
17. Any surgical procedure in the treatment area within the last six months or before complete healing.
18. Treating over tattoo or permanent makeup.
19. Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.
20. As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gronski, Study Director — Venus Concept
Locations (1):
- Sadick Research Group, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 20
Completed | 14
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Subject Satisfaction
Description: Subjects' assessment of satisfaction with the treatment using a 5-point Subject Satisfaction Scale at 12 weeks post-treatment. The Subject Satisfaction Scale is a five-grade subjective test. Possible responses were (4) Very Satisfied, (3) Satisfied, (2) Having No Opinion, (1) Unsatisfied, and (0) Very Unsatisfied.
Time Frame: 12 Weeks Post-Final Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 10
units on a scale | 3.5 (0.5)

2. Secondary Outcome: Treatment Pain
Description: Subject's assessment of discomfort and pain assessed immediately after treatments as measured by a 10 cm visual analog scale (VAS). The Visual Analog Scale is a scale from 0 cm (no pain) and 10 cm (pain as bad as it can be).
Time Frame: Average of all treatments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 20
units on a scale | 4.2 (1.7)

3. Secondary Outcome: Subject Scale - 5 Point Scale for Treatment Tolerability
Description: Subject's assessment of treatment tolerability as measured by a 5 point scale. Participants were asked about their treatment tolerability level immediately post-treatment. Possible scores were; (4) Very Tolerable, (3) Tolerable, (2) Having No Opinion, (1) Intolerable, and (0) Very Intolerable.
Time Frame: Average of all treatments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 20
units on a scale | 3.1 (0.4)

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=20)
Trauma on chin (Skin and subcutaneous tissue disorders) | 1 (1)
Trauma on forehead (Skin and subcutaneous tissue disorders) | 1 (1)
Acne and new scars (Skin and subcutaneous tissue disorders) | 1 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT04827680/Prot_SAP_000.pdf